CLINICAL TRIAL: NCT03272646
Title: The Naples Prognostic Score in Gastric Cancer Patients Undergoing Surgery
Brief Title: Prognostic Performance of the Naples Prognostic Score
Acronym: NPS
Status: Completed | Type: Observational
Sponsor: University of Campania Luigi Vanvitelli (Other)
Responsible Party: Principal Investigator, Gennaro Galizia, Full Professor of Surgery, University of Campania Luigi Vanvitelli
Other Study IDs: UNI Naples Vanvitelli
Record Dates: First submitted 2017-09-01; First posted 2017-09-05 (Actual); Last update posted 2017-09-05 (Actual); Status verified 2017-09

CONDITIONS: Nutritional and Metabolic Diseases; Oncologic Disorders
Keywords: Gastric Cancer
MeSH Terms: conditions — Nutritional and Metabolic Diseases; Stomach Neoplasms | interventions — Surgical Procedures, Operative

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 17 Years
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Group 1 or NPS = 0: Patients undergoing surgery without alterations of the albumin and cholesterol levels, with normal NLR and LMR ratios.
  Interventions: Procedure: surgery
- Group 2 or NPS >0 and < 3: Patients undergoing surgery with NPS between 1 or 2
  Interventions: Procedure: surgery
- Group 3 or NPS > 2: Patients undergoing surgery with three or four alterations
  Interventions: Procedure: surgery

INTERVENTIONS:
Procedure: surgery — gastric resection or total gastrectomy
  Other Names: radical surgery

SUMMARY:
To investigate the prognostic performance of the Naples Prognostic Score in gastric cancer patients undergoing surgery

DETAILED DESCRIPTION:
The outcome of oncological patients is related not only to the tumor status but also to the host. Particularly the patient's immune and nutritional status have been recently associated with short- and long-term outcome in gastric and other cancers. In addition, there is growing evidence that systemic inflammation plays a crucial role in the carcinogenesis and progression of gastric cancer. The neutrophil to lymphocyte ratio (NLR), and, more recently, the lymphocyte to monocyte ratio (LMR) have been shown to be independently correlated with prognosis in patients with gastric cancer who underwent surgery, and preoperative albumin and cholesterol levels seem to be adequate mirrors of the nutritional status of the host.

The investigators have already demonstrated that a new scoring system, which they called Naples prognostic score (NPS), based on a composite score of albumin and cholesterol concentrations, along with NLR and LMR is a simple tool strongly associated with long-term outcome in patients undergoing surgery for colorectal cancer.

The aim of this study is to assess the correlation between the NPS and clinicopathological characteristics, postoperative complication rate and long-term outcome in patients undergoing surgery for gastric cancer. Furthermore, the new prognostic scoring system will be compared with previously developed ones and the current TNM staging system to evaluate its performance.

All patients who underwent surgery for proven gastric adenocarcinoma at the Division of Surgical Oncology of the Gastrointestinal Tract of the University of Campania (Naples, Italy), from January 2000 to December 2015 will be enrolled in the present study.

ELIGIBILITY:
Inclusion Criteria:

* all patients undergoing surgery at our institution for proven gastric adenocarcinoma will be enrolled in the present study

Exclusion Criteria:

* Patients with lower esophageal adenocarcinoma or cancer crossing the esophagogastric junction with its epicenter in the proximal 2 cm of stomach, which were taken apart from stomach cancers in the last two AJCC cancer staging editions, will be excluded.
* Patients with ongoing infections, concomitant immune-mediated diseases, or on drugs capable of affecting neutrophil and/or lymphocyte counts (e.g., steroids, immunosuppressants, etc.) will be excluded from the study.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with proven gastric adenocarcinoma undergoing surgery.
Sampling Method: Non-Probability Sample
Enrollment: 477 (Actual)
Dates: Start 2000-01-01 (Actual); Primary Completion 2015-12-31 (Actual); Study Completion 2017-06-30 (Actual)

PRIMARY OUTCOMES:
Prognostic performance of NPS. | through study completion, an average of 1 year
  Corrlation between preoperative NPS and outcome (i.e. overall survival in all patients, and disease-free survival in radically resected patients). The prognostic performance of NPS will be compared to that of the prognostic nutritional index (PNI), the controlling nutritional status (CONUT) score, the systemic inflammation score (SIS), and the TNM staging system.

CONTACTS AND LOCATIONS:
Overall Officials: Gennaro Galizia, MD, Principal Investigator — University of Campania 'Luigi Vanvitelli'

IPD SHARING:
Plan to Share IPD: Yes
All data will be made available by contacting the principal investigator.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: at the end of the study
Access Criteria: gennaro.galizia@unicampania.it